CLINICAL TRIAL: NCT01964599
Title: Potato Fiber and Gastrointestinal Function: Phase 3 (Grant #94521)
Brief Title: Potato Fiber and Gastrointestinal Function: Phase 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 215-2011
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Gastrointestinal Symptoms; Gastrointestinal Transit Time; Stool Frequency
Keywords: Fiber; Gastrointestinal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-RS (Other): 14 days consuming the PF-RS containing 30 g fiber and then 14 days consuming the control containing no fiber
  Interventions: Dietary Supplement: PF-RS; Dietary Supplement: Control
- PF-RO1 (Other): 14 days consuming the PF-RO1 containing 30 g fiber and then 14 days consuming the control containing no fiber
  Interventions: Dietary Supplement: PF-RO1; Dietary Supplement: Control
- PF-RO2 (Other): 14 days consuming the PF-RO2 containing 30 g fiber and then 14 days consuming the control containing no fiber
  Interventions: Dietary Supplement: PF-RO2; Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: PF-RS — n=20 will consume PF-RS containing 30 g potato fiber for 14 days and will consume a control containing no fiber for 14 days.
  Arms: PF-RS
Dietary Supplement: PF-RO1 — n=20 will consume PF-RO1 containing 30 g potato fiber for 14 days and will consume a control containing no fiber for 14 days.
  Arms: PF-RO1
Dietary Supplement: PF-RO2 — n=20 will consume PF-RO2 containing 30 g potato fiber for 14 days and then will consume a control containing no fiber for 14 days.
  Arms: PF-RO2
Dietary Supplement: Control

SUMMARY:
The primary physiological impacts of fiber intake include the gastrointestinal effects of stool bulking, increased stool frequency and decreased gastrointestinal transit time (GTT). Fermentation of resistant starches by microbiota increases bacterial numbers, which increases fecal bulk and may impact frequency and transit time. The purpose of this study is to determine the effects of resistant potato starches (potato fiber) on stool frequency, transit time and microbiota in healthy individuals.

DETAILED DESCRIPTION:
Potato fiber (PF-RS, PF-RO1 and PF-RO2), supplemented in the diet of healthy individuals (n=60; 20 per group) and providing 30 g per day of fiber, will result in a significant changes in gastrointestinal function and microbiota profile.

Objectives:

1. To determine the effect of potato fibers on stool frequency, gastrointestinal transit time and gastrointestinal symptoms.
2. To determine the effect of potato fibers on microbial diversity in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* must be between the ages of 18 and 65.
* must be willing to complete daily questionnaires.
* must be willing to provide a social security number to receive study payment. Note: the subject can still participate if unwilling to provide SS#, but no financial reimbursement can be provided.
* must have internet access for the duration of the study
* must have usual fiber intake of <20 g/d based on Food Frequency Questionnaire such as the Block Fruit/Vegetable/Fiber Screener
* must be willing to consume kool-aid everyday for 2 periods of 14 days
* must be willing to provide stool samples

Exclusion Criteria:

* must not have a physician-diagnosed gastrointestinal disease or condition (such as ulcerative colitis, Crohn's disease, gastroparesis, cancer, peptic ulcer disease, Celiac disease, short bowel disease, ileostomy, colostomy other than GERD, constipation, diverticular disease)
* must not have a food allergy
* must not take dietary supplements (prebiotic and fiber supplements)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Stool Frequency | 6 weeks
  Change in stool frequency determined by the daily questionnaire

SECONDARY OUTCOMES:
Gastrointestinal transit time | 6 weeks
  Change in gastrointestinal transit time determined by the Bristol Stool Scale
Gastrointestinal symptoms | 6 weeks
  Change in gastrointestinal symptoms determined by the daily questionnaire
Microbial diversity | 6 weeks
  Baseline, treatment, control and washout stools (for a total of 6 samples) for each subject will be sampled for DNA isolation for microbiota studies. Microbial diversity measured by DGGE profiling (detects large distortions), qPCR to quantify changes and 16S rRNA sequencing (454) to identify treatment effects on specific bacteria (discovery) will be undertaken.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Dahl, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Food Science & Human Nutrition Dept, Gainesville, Florida, United States